CLINICAL TRIAL: NCT04908410
Title: The Norwegian Addiction, Pain and Trauma Study
Acronym: NOR-APT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); Norwegian Center for Violence and Traumatic Stress Studies (Other); The Hospital of Vestfold (Other); Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Ingeborg Skjarvo, Researcher, University Hospital, Akershus
Other Study IDs: 2020/173249(REK)
Record Dates: First submitted 2021-05-18; First posted 2021-06-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Post-traumatic Stress Disorder; Substance Use Disorders
Keywords: Opioid; Alcohol; Amphetamine; Cannabis; Marijuana; Methadone; Buprenorphine; Opioid maintenance treatment; Chronic pain; Post-traumatic stress
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In populations with substance use disorders (SUD), there is a high prevalence of chronic pain with various underlying causes. Chronic pain can complicate the treatment of SUD and lead to poorer treatment outcomes. There is a need for a better understanding of the connections and interactions between chronic pain and substance use and dependence.

Further, there is a high prevalence of chronic pain among patients with post-traumatic stress disorder (PTSD). As there is an overlap between populations with SUD and PTSD, taking potentially traumatizing life-experiences and post-traumatic stress symptoms into account can provide a better understanding of chronic pain in populations with SUD.

The Nor-APT study is a cross-sectional study, recruiting from outpatient and inpatient substance use treatment centres connected to four hospitals. Participants complete a questionnaire about substance/medication use, pain and how pain affect function, stressful life events and post-traumatic stress symptoms. Patients can consent to self-reported data being linked to retrospective and prospective longitudinal data from national demographic and health registries.

The purpose of the study is to contribute to a better understanding and treatment of chronic pain among people with substance use disorders (SUD), and to contribute to the understanding of co-occurring substance use, chronic pain and post-traumatic stress symptoms.

The over-arching research aims are to:

I. Describe the prevalence and characteristics of pain for people in need of treatment for substance/medication use/dependence.

II. Describe how the pain affects physical and emotional functioning, and subjective quality of life.

III. Explore any connections between substance/medication use and pain, both what came first and any ways substance/medication use and pain affect each other.

IV. Explore the connection between chronic pain, potentially traumatizing life events and post-traumatic stress symptoms.

V. Explore how treatments received and how treatment affects outcomes.

In addition, we will explore whether participants' experiences can be categorized into typical trajectories for how substance use, chronic pain and stressful life events occur and develop over the life span.

DETAILED DESCRIPTION:
INTRODUCTION

Chronic pain and substance use

The prevalence of chronic pain is high among persons with opioid dependence and alcohol dependence. According to a recent review, it is common for patients to use both opioids and alcohol, and this is seen especially in cases where the patient also experiences chronic pain. Nevertheless, alcohol use is often omitted from research on opioids and chronic pain. The review concludes that there is a great need for more knowledge about co-use of alcohol and opioids in people with chronic pain.

The high prevalence of chronic pain in populations with opioid or alcohol dependence could be related to comorbid physical illness and injuries, which is prevalent among opioid dependent patients. It is also possible that use of opioids or alcohol can contribute to pain sensitivity and worsening of pain over time.

There have been few studies focusing on chronic pain and dependence on other substances than opioids or alcohol. The prevalence of chronic pain among people with, for example, amphetamine dependence or cannabis dependence has received little attention, although cannabinoids are also used as prescription painkillers.

A study of the general population in the United States found a link between chronic pain and marijuana use, but could not discern whether the pain or marijuana use came first. In a small study, two out of five people using marijuana or cocaine reported using the substances as pain relief. Amphetamine is also a highly relevant substance when it comes to pain, as amphetamines can be analgesic, and can enhance the analgesic effect of opioids.

Chronic pain is associated with poorer treatment outcomes, however there is little knowledge about how co-occurring chronic pain and substance dependence develops over time. More knowledge about the mechanisms behind co-occurring chronic pain and dependence can contribute to better treatment options for patients, both when it comes to the treatment of pain and dependence.

Chronic pain and PTSD

Chronic pain and pain intensity have a documented association with post-traumatic stress disorder (PTSD) in the general population, but have not been much explored among people with dependence. A small study has found a higher prevalence of chronic pain among people with co-occurring substance dependence and PTSD, but the study was not large enough (n = 133) to distinguish between dependence on different types of substances. One study (n = 150) found a higher prevalence of PTSD among methadone patients with chronic pain.

Unfortunately, PTSD is a diagnosis that has historically been considered difficult to treat among people with substance use disorder. Therefore PTSD is undertreated for these patients.

The link between chronic pain and PTSD is not fully understood. In some cases, the pain may be caused by a physical injury in connection with the event that caused the PTSD. Beyond these cases, some theories focus on shared vulnerability, or that chronic pain and PTSD reinforce each other through excessive reactions to or misinterpretation of stress or pain stimuli. Other theories focus on the biological aspects, such as dysregulation of the nervous system or dysregulation of opioid receptors.

It is also possible that the PTSD symptoms associated with overactivation may drive the association between PTSD and pain. This makes it relevant to explore any potential interaction effects of PTSD symptoms and the use of sedative and stimulating substances/medications on the experience of pain.

A better understanding of the links between chronic pain, PTSD and dependence can mean a lot for better treatment of patients with comorbid substance dependence, PTSD and pain disorders.

METHODS

Design. Cross-sectional survey study, with linkage to retrospective and prospective registry data. The NOR-APT study employs a rarely utilized research design where survey data containing the patients' self-reported experiences are combined with high quality, nearly complete, longitudinal registry data from the first and second line health care services and the prescription database, as well as sociodemographic registries.

Data from the first registration of the patient in the registries can be linked to self-reported data through personal identification numbers retained by all residents, providing a complete history of treatments and diagnoses.

It is a multicentre study, with data collected from over 20 substance use treatment centres in the catchment areas for Akershus University Hospital, Oslo University Hospital, Vestfold Hospital Trust and Telemark Hospital in Norway.

Participants. The goal is to recruit 1 500 patients entering any form of substance use treatment at the 20+ collaborating inpatient and outpatient clinics.

Staff at the treatment centres are instructed to ask all patients. At the time-points where 500 and 1 000 questionnaires have been completed, the investigators will assess the distribution of participants according to their primary substance use problem/the substance they are in treatment for. If the distribution is skewed in a manner that may not give enough data about some sub-groups of substance users, the investigators may encourage staff at the treatment centres to continue with more selective recruitment of the patient groups that are underrepresented. For instance, many patients are treated for opioid or alcohol dependence, so this group may be recruited faster and more easily, while patients with a primary dependence to cannabis or amphetamines may be fewer and could require more time and effort to reach a sufficiently large sample size.

Materials. The questionnaire was developed based on the research questions, previous literature, and in collaboration with the clinicians that see the patient groups in their day to day practice at Akershus University Hospital and Oslo University Hospital. The questionnaire was piloted on 10 patients with different substance use patterns, where patients were asked to comment on the experience of filling in the questionnaire, the length and clarity of the questions, and give any other comments or suggestions. Further adjustments to the layout and wording of certain questions were made based on the results of the piloting.

To make the data-collection process as uniform as possible, a questionnaire guide for staff was made, with a standard text for introducing and explaining the questionnaire to patients, and with a walk-through of the questions with additional explanations, definitions and problem-solving for common issues when filling out the different type of questions. In the guide, other topics related to collecting survey-data were also addressed, such as concerns related to missing responses for data validity and how to balance the preference for complete answers with ensuring that all questions were answered on a completely voluntary basis.

An instructional 15 minute video for staff was made, with an explanation of the background and purpose of the study, as a measure to increase understanding and motivation for recruiting patients to the study.

Registry data: The Norwegian registries consist of high-quality data on for instance treatment episodes, diagnoses, prescribed medications and socioeconomic variables, with nearly complete data for all individuals in Norway.

Procedure. Each treatment centre has a study coordinator responsible for ensuring all staff has access to questionnaires, guides and the instructional video. The coordinators task is to inform staff and distributed the study material. The coordinator will also report on progress, issues and concerns to the central study coordinators throughout the data collection period.

Staff at the treatment centres are instructed to invite all patients (except those affected by the exclusion criteria) to participate. Patients will be informed that participation is voluntary and that declining to participate will not affect the treatment they receive, about the purpose of the study and how the information they give will be handled. The number of patients that decline participation will be logged, and if the patients consent to disclosing the information, the gender, age and which substance they are in treatment for/their primary substance problem, will also be logged for patients that decline participation.

Patients that agree to participate will complete the consent form and the questionnaire. If they wish to withdraw from the study at a later time, they can contact the treatment centre or the research group.

For participants who consent to linkage of questionnaire data with longitudinal registry data, linkage to retrospective registry data will be performed about a year after collection of questionnaire data has been completed, and linkage to prospective registry data will be done 5-6 years after the collection of questionnaire data have been completed. Linkages are performed by the Norwegian Institute of Public Health and Statistics Norway, based on the patients explicit consent and unique personal identification number.

ELIGIBILITY:
Inclusion Criteria:

* Patient in substance use treatment at a treatment centre under Akershus University Hospital, Oslo University Hospital, Vestfold Hospital or Telemark Hospital.

Exclusion Criteria:

Staff considers the patient to be unable to give informed consent/valid responses on the questionnaire OR staff considers participation to be too stressful/burdensome to the patient. Staff are asked to take the following into consideration when making their assessment:

* Acute withdrawal
* Acute intoxication
* Serious mental health concerns
* Serious physical health concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (ages 18 years - unlimited) in treatment for substance use disorders at outpatient and inpatient treatment centers connected to Akerhus University Hospital or Oslo University Hospital, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic pain (ICD-10) | T1 (at enrollment in study)
  Defined as having experienced pain with a duration of at least 3 months.
European-Addiction Severity Index (EuropASI), Section E | T1 (at enrollment in study)
  * Types of substances used (life-time), age of first use, and frequency of use in the last 4 weeks.
  * Intravenous use (life-time and last 4 weeks)
  Modifications:
  1. We updated the list of substances to better match the relevant substances in use today: Alcohol to intoxication; OMT medications (methadone; subutex; suboxone); Other opioid painkillers (e.g. morphine, oxycodone, tramadol); Cannabis; Amphetamine/ Methamphetamine; Cocaine; Benzodiazepines; GHB; Hallucinogenics (e.g. LSD, mushrooms, mescaline); Anabolic steroids; Khat.
  2. Frequency of use in the last 4 weeks: the response categories "used not more than 2-3 times per month" and " used 1-3 times a week" were collapsed into one category "used a few times", leaving three categories: "Not used", "used a few times" and "every day/nearly every day".
The Stressful Life-Events Screening Questionnaire (SLESQ) | T1 (at enrollment in study)
  The SLESQ assesses exposure to stressful life-events (yes/no) that could be potentially traumatizing. This version has been shortened and adapted in previous studies at the Norwegian Centre for Violence and Traumatic Stress Studies (NKVTS) for use in Norway and includes a list of 15 types of stressful events. This variable will be used to assess the prevalence of different types of stressful life-events. In addition the number of events can be summed to indicate the extent of exposure to stressful life-event, with a range from 0 events to 15.
  Modifications:
  1. Two events have been added: Being directly involved in a natural disaster and having been repeatedly ridiculed, put down, ignored or told you were no good by someone outside the family.
  2. When several of the 15 types of events have occured, the participants' age at the time of the event is only recorded for the first event and the event that gives the participant the most symptoms now.
The PTSD Checklist for DSM-5 - short version (PCL-5 short) | T1 (at enrollment in study)
  The short version of the PTSD Checklist for DSM-5 includes 4 items: 1 item for each symptom cluster for the diagnosis of PTSD according to the DSM-5.
  Participants indicate how much each symptom has bothered them in the last month on a scale from 0 to 4 ("Not at all" to "Very much"). The sum score ranges from 0 to 16. A score above the cut score of 10 indicates risk for PTSD, and has previously been validated as a diagnostic indicator.

SECONDARY OUTCOMES:
Pain characteristics | T1 (at enrollment in study)
  Patients that report any pain in the last 4 weeks are asked:
  * to indicate the location/s of the pain on a body map with 25 different pain locations (from the Norwegian Pain Association)
  * to indicate any generalized pain in the skin, muscles, joints or skeleton/bones (selfmade checklist).
  * the duration of their pain (less than 3 months; 3-12 months; 1-3 years; 4-6 years; 7-10 years; more than 10 years)
  * the cause of their pain (illness; accident/injury; violence; surgery; other; unknown), their age at that time and whether they believe the cause was related to their substance use (selfmade questions, the list of causes collected from previous studies).
The Brief Pain Inventory: Pain intensity | T1 (at enrollment in study)
  Pain intensity will be assess with 4 items addressing pain intensity right now; on average; the strongest in the last week; the weakest in the last week. Responses are given on an 11 point numeric rating scale from 0 "No pain" to 10 "The worst pain imaginable". These 4 items can be used independently or averaged.
The Brief Pain Inventory: Pain interference | T1 (at enrollment in study)
  Pain interference on different life domains in the last week will be assessed with 7 items from the BPI: general activity, ability to walk, normal work/housework, mood, sleep, relationships to others, enjoyment of life
  Responses are given on an 11 point numeric rating scale from 0 "Not influenced at all" to 10 "Completely influenced".
  The 7 items can be averaged to give an overall interference score from 0 (low) to 10 (high), or they can be divided into affective interference (mood, sleep, relationships, enjoyment of life) and activity interference (walking, activity, work).
  In addition, we include1 selfmade item in the same format, about interference on subjective quality of life: satisfaction with life.
Other pain related questions (selfmade) | T1 (at enrollment in study)
  * Have you contacted a medical doctor for help with your pain? (Yes/no). If yes, age at the time (open ended question)
  * Did you receive treatment for your pain? (yes/no) If yes, what type of treatment (open ended question).
  * Is it difficult for you now to stop using substances/medications because of
  * pain? (No/ A little/ Very)
  * worrying about pain? (No/ A little/ Very)
  * Are there substance/medications (including over the counter pain medications) that...
  * ...help with your pain? (open ended question)
  * ... make your pain worse? (open ended question)
  * The first time you used opioids, was it to relieve pain? (Never used opioids/No/Yes/Don't know)
  * Has pain ever influenced the type of medication received in OMT? (No/Yes/Don't know) If yes, which medication? (open ended), what was your age at the time? (open ended), Any comments? (open ended).
Opioid maintenance treatment (OMT) history (selfmade) | T1 (at enrollment in study)
  * Have you ever been in OMT? (No/Methadone/Subutex/Buvidal/Suboxone/Other (specify)) Age at the time of the first prescription.
  * Are you in OMT now? (No/Methadone/Subutex/Buvidal/Suboxone/Other (specify)) Age at the start of this prescription.
Subjective quality of life (QOL-1) | T1 (at enrollment in study)
  - How satisfied are you with your life? The response is given on an 11-point numeric rating scale, from 0 "Not satisfied at all" to 10 "Very satisfied".
Demographics | T1 (at enrollment in study)
  * Age
  * Gender (Woman/man)
  * Are you currently working/studying? (No/Yes (full or parttime) OR On sickleave/Retired/Disabled)
Nicotine use | T1 (at enrollment in study)
  * Do you smoke cigarettes or a pipe? (Yes/No)
  * Do you use snuff? (Yes/No)
ICD-10/11 diagnostic codes | Retrospective (back to 2008) and prospective (5 year follow-up from completion of the questionnaire)
  From the Norwegian Patient Registry (NPR) we wi receive all registered contacts/treatments with the secondary specialist health care services (for somatic diseases, mental health and substance dependence), including ICD codes and dates for treatment start and end.
Prescribed medications | Retrospective (back to 2004) and prospective (5 year follow-up from completion of the questionnaire)
  From the Norwegian Prescription Database (NorPD) we will receive all registered medications with dates for when they were collected from the pharmacy.
Treatments in the primary health services | Retrospective (back to 2016) and prospective (5 year follow-up from completion of the questionnaire)
  From the municipal health registry (KPR) we will receive codes for all treatments in the primary (municipal) health services, including emergency care, general practitioners and dentists.
Pain treatment | Retrospective (back to 2013) and prospective (5 year follow-up from completion of the questionnaire)
  From the national quality registry for pain treatment (SmerteReg) we can receive additional details concerning pain treatment
Treatments of patients with severe physical trauma | Retrospective (since establishment of database) and prospective (5 year follow-up from completion of the questionnaire)
  From the national traumaregister (NTR) we can receive information on patients who have received treatments for severe physical trauma.
Cancer diagnosis and treatments | Retrospective (since establishment of database) and prospective (5 year follow-up from completion of the questionnaire)
  From the Cancer registry we can receive additional information on cancer diagnosis and treatments.
Time and cause of death | Prospective (5 year follow-up from completion of the questionnaire)
  From the Cause of death registry we will receive the date and cause of death for patients who have died during the 5-year follow-up period.
Level of education | Retrospective (back to 1960s) and prospective (5 year follow-up from completion of the questionnaire)
  From the demographic database of Statistics Norway we will receive information on the highest level of completed education.
Birthcountry and immigration status | Retrospective (back to 1960s) and prospective (5 year follow-up from completion of the questionnaire)
  From the demographic database of Statistics Norway we will receive information on birth country and 1st, 2nd and 3rd generation immigration status.
Income and employment status | Retrospective (back to 1960s) and prospective (5 year follow-up from completion of the questionnaire)
  From the demographic database of Statistics Norway we will receive information of types of income and employment status, sick-leave and benefits.
Living conditions | Retrospective (back to 1960s) and prospective (5 year follow-up from completion of the questionnaire)
  From the demographic database of Statistics Norway we will receive information on type of dwelling, number of persons in the household, moves between houses.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Skjærvø, PhD, Principal Investigator — Ingeborg Skjærvø
Locations (4):
- Norway (4):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Telemark Hospital, Skien
  - The Hospital in Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Latif ZH, Skjaervo I, Solli KK, Tanum L. Chronic Pain Among Patients With an Opioid Use Disorder. Am J Addict. 2021 Jul;30(4):366-375. doi: 10.1111/ajad.13153. Epub 2021 Mar 19. PMID 33738870
- [Background] Rosenblum A, Joseph H, Fong C, Kipnis S, Cleland C, Portenoy RK. Prevalence and characteristics of chronic pain among chemically dependent patients in methadone maintenance and residential treatment facilities. JAMA. 2003 May 14;289(18):2370-8. doi: 10.1001/jama.289.18.2370. PMID 12746360
- [Background] Boissoneault J, Lewis B, Nixon SJ. Characterizing chronic pain and alcohol use trajectory among treatment-seeking alcoholics. Alcohol. 2019 Mar;75:47-54. doi: 10.1016/j.alcohol.2018.05.009. Epub 2018 May 25. PMID 30359794
- [Background] Witkiewitz K, Vowles KE. Alcohol and Opioid Use, Co-Use, and Chronic Pain in the Context of the Opioid Epidemic: A Critical Review. Alcohol Clin Exp Res. 2018 Mar;42(3):478-488. doi: 10.1111/acer.13594. Epub 2018 Feb 6. PMID 29314075
- [Background] Larney S, Peacock A, Mathers BM, Hickman M, Degenhardt L. A systematic review of injecting-related injury and disease among people who inject drugs. Drug Alcohol Depend. 2017 Feb 1;171:39-49. doi: 10.1016/j.drugalcdep.2016.11.029. Epub 2016 Dec 8. PMID 28013096
- [Background] Pud D, Cohen D, Lawental E, Eisenberg E. Opioids and abnormal pain perception: New evidence from a study of chronic opioid addicts and healthy subjects. Drug Alcohol Depend. 2006 May 20;82(3):218-23. doi: 10.1016/j.drugalcdep.2005.09.007. Epub 2005 Oct 17. PMID 16229972
- [Background] Phillips K, Clauw DJ. Central pain mechanisms in chronic pain states--maybe it is all in their head. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):141-54. doi: 10.1016/j.berh.2011.02.005. PMID 22094191
- [Background] Egli M, Koob GF, Edwards S. Alcohol dependence as a chronic pain disorder. Neurosci Biobehav Rev. 2012 Nov;36(10):2179-92. doi: 10.1016/j.neubiorev.2012.07.010. Epub 2012 Sep 11. PMID 22975446
- [Background] Apkarian AV, Neugebauer V, Koob G, Edwards S, Levine JD, Ferrari L, Egli M, Regunathan S. Neural mechanisms of pain and alcohol dependence. Pharmacol Biochem Behav. 2013 Nov;112:34-41. doi: 10.1016/j.pbb.2013.09.008. Epub 2013 Oct 2. PMID 24095683
- [Background] Hill KP. Medical Marijuana for Treatment of Chronic Pain and Other Medical and Psychiatric Problems: A Clinical Review. JAMA. 2015 Jun 23-30;313(24):2474-83. doi: 10.1001/jama.2015.6199. PMID 26103031
- [Background] Zvolensky MJ, Cougle JR, Bonn-Miller MO, Norberg MM, Johnson K, Kosiba J, Asmundson GJ. Chronic pain and marijuana use among a nationally representative sample of adults. Am J Addict. 2011 Nov-Dec;20(6):538-42. doi: 10.1111/j.1521-0391.2011.00176.x. Epub 2011 Oct 4. PMID 21999500
- [Background] Alford DP, German JS, Samet JH, Cheng DM, Lloyd-Travaglini CA, Saitz R. Primary Care Patients with Drug Use Report Chronic Pain and Self-Medicate with Alcohol and Other Drugs. J Gen Intern Med. 2016 May;31(5):486-91. doi: 10.1007/s11606-016-3586-5. Epub 2016 Jan 25. PMID 26809204
- [Background] Chen AL, Chen TJ, Waite RL, Reinking J, Tung HL, Rhoades P, Downs BW, Braverman E, Braverman D, Kerner M, Blum SH, DiNubile N, Smith D, Oscar-Berman M, Prihoda TJ, Floyd JB, O'Brien D, Liu HH, Blum K. Hypothesizing that brain reward circuitry genes are genetic antecedents of pain sensitivity and critical diagnostic and pharmacogenomic treatment targets for chronic pain conditions. Med Hypotheses. 2009 Jan;72(1):14-22. doi: 10.1016/j.mehy.2008.07.059. Epub 2008 Oct 31. PMID 18951726
- [Background] Larson MJ, Paasche-Orlow M, Cheng DM, Lloyd-Travaglini C, Saitz R, Samet JH. Persistent pain is associated with substance use after detoxification: a prospective cohort analysis. Addiction. 2007 May;102(5):752-60. doi: 10.1111/j.1360-0443.2007.01759.x. PMID 17506152
- [Background] Sharp TJ, Harvey AG. Chronic pain and posttraumatic stress disorder: mutual maintenance? Clin Psychol Rev. 2001 Aug;21(6):857-77. doi: 10.1016/s0272-7358(00)00071-4. PMID 11497210
- [Background] Fishbain DA, Pulikal A, Lewis JE, Gao J. Chronic Pain Types Differ in Their Reported Prevalence of Post -Traumatic Stress Disorder (PTSD) and There Is Consistent Evidence That Chronic Pain Is Associated with PTSD: An Evidence-Based Structured Systematic Review. Pain Med. 2017 Apr 1;18(4):711-735. doi: 10.1093/pm/pnw065. PMID 27188666
- [Background] Moeller-Bertram T, Keltner J, Strigo IA. Pain and post traumatic stress disorder - review of clinical and experimental evidence. Neuropharmacology. 2012 Feb;62(2):586-97. doi: 10.1016/j.neuropharm.2011.04.028. Epub 2011 May 10. PMID 21586297
- [Background] Ouimette P, Goodwin E, Brown PJ. Health and well being of substance use disorder patients with and without posttraumatic stress disorder. Addict Behav. 2006 Aug;31(8):1415-23. doi: 10.1016/j.addbeh.2005.11.010. Epub 2005 Dec 27. PMID 16380217
- [Background] Barry DT, Beitel M, Cutter CJ, Garnet B, Joshi D, Rosenblum A, Schottenfeld RS. Exploring relations among traumatic, posttraumatic, and physical pain experiences in methadone-maintained patients. J Pain. 2011 Jan;12(1):22-8. doi: 10.1016/j.jpain.2010.04.006. Epub 2010 Jun 20. PMID 20646965
- [Background] Flanagan JC, Korte KJ, Killeen TK, Back SE. Concurrent Treatment of Substance Use and PTSD. Curr Psychiatry Rep. 2016 Aug;18(8):70. doi: 10.1007/s11920-016-0709-y. PMID 27278509
- [Background] Pacella ML, Girard JM, Wright AGC, Suffoletto B, Callaway CW. The Association Between Daily Posttraumatic Stress Symptoms and Pain Over the First 14 Days After Injury: An Experience Sampling Study. Acad Emerg Med. 2018 Aug;25(8):844-855. doi: 10.1111/acem.13406. PMID 29513381
- [Derived] Skjaervo I, Marciuch A, Digranes LW, Folleras LM, Mordal J, Solli KK, Abel EKF, Amundsen K, Egeland K, Haugen BK, Holmoy B, Skoftedalen JG, Weimand BM, Tanum L. Chronic Pain and Posttraumatic Stress Among Patients in Substance Use Treatment: Protocol for NOR-APT, a Longitudinal Cohort Study. JMIR Res Protoc. 2025 Dec 24;14:e67663. doi: 10.2196/67663. PMID 41442162

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04908410/SAP_000.pdf